CLINICAL TRIAL: NCT03517202
Title: Duration of Stay for Outpatient Surgery After Tension Free Vaginal Tape (TVT) Urologic Surgery : Neuraxial Versus General Anesthesia
Brief Title: Duration of Stay After Urologic Surgery : Neuraxial Versus General Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7001
Record Dates: First submitted 2018-04-24; First posted 2018-05-07 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-03

CONDITIONS: Urinary Retention
Keywords: Urologic surgery; Urinary incontinence; Tension Free Vaginal Tape; Post-operative urinary retention; Outpatient surgery
MeSH Terms: conditions — Urinary Retention; Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Outpatient midurethral surgery is a frequent surgery. It is performed either under general anesthesia or neuraxial anesthesia. A frequent complication is postoperative urinary retention requiring urinary catheterization, which implies a higher infectious risk.

The investigators compared the complication rate after TVT surgery depending on the type of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Sex: Female
* Patient who has consented to the use of her medical data for research purposes.
* Patient undergoing outpatient urinary incontinence surgery using TVT between 2012 and 2016

Exclusion Criteria:

* Specific clinical forms of the disease,
* Interfering treatments and associated diseases, history,
* Refusal of the patient to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient undergoing outpatient urinary incontinence surgery using TVT between 2012 and 2016
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2018-03-13 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
The investigators compared the rate of complications after TVT surgery depending on the type of anesthesia and the need for urinary catheterization, requiring longer hospital stay after surgery. | The period from January 1st, 2012 to December 31st, 2016 will be examined
  Patients hospitalized at Strasbourg University Hospital from 2012 to 2016.

CONTACTS AND LOCATIONS:
Overall Officials: Valentina FAITOT, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Service d'Anesthésiologie - Réanimation, Strasbourg, France